CLINICAL TRIAL: NCT05810883
Title: Prevalence and Risk Factors of Insulin Resistance in Overweight and Obese Adolescents
Brief Title: Prevalence of IR in Overweight and Obese Adolescents
Acronym: IR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yara Mostafa, Pediatric Resident Physician, Assiut University
Other Study IDs: IR in Overweight Adolescents
Record Dates: First submitted 2022-04-12; First posted 2023-04-13 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Hematologic Tests; Waist Circumference

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood tests include Serum Fasting Insulin and Serum Blood Glucose, along with lipid profile
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Insulin Resistant Group: HOMA-IR score of ≥ 3.4
  Interventions: Diagnostic Test: Blood Tests; Serum Fasting Insulin and Glucose
- Non-Insulin Resistant: HOMA-IR score of less than 3.4
  Interventions: Diagnostic Test: Blood Tests; Serum Fasting Insulin and Glucose

INTERVENTIONS:
Diagnostic Test: Blood Tests; Serum Fasting Insulin and Glucose — Laboratory results of blood samples, for high-density lipoprotein (HDL), low-density protein (LDL), triglycerides, and total cholesterol (TC) will be evaluated for this study. Fasting Insulin and fasting glucose levels will be used to calculate IR.
  Insulin Resistance will be calculated using Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) (FPG (mmol/L) × FPI (mU/L)/22.5) [21] and defined as HOMA-IR ≥ 3.4
  Other Names: Anthropometric Measurements including BMI and Waist circumference

SUMMARY:
The aim of this study is to determine the prevalence of Insulin Resistance (IR) among overweight and obese adolescents using HOMA-IR scores and identify lifestyle risk factors in the IR and Non-IR group.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents of ages ≥ 10-≤18 years, of both sexes who are Overweight (BMI > 85th percentile) or Obese (BMI > 95th percentile).

Exclusion Criteria:

* Obesity due to Secondary causes as Cushing disease or hypothyroid patients, and any other patients with Chronic illness.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescent Children attending Hospital or Primary care clinics in Egypt whom fit the criteria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-05-11 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants of the Obese or Overweight category with elevated Serum Fasting Insulin and Serum Fasting glucose scores | Baseline
  Measuring Serum Fasting Insulin and Fasting Glucose levels to calculate HOMA-IR scores Insulin Resistance will be calculated using Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) (Fasting Plasma Glucose (mmol/L) × Fasting Plasma Insulin (mU/L)/22.5) and defined as HOMA-IR ≥ 3.4 to Detect Prevalence of IR, higher scores indicating increased Insulin Resistance.

SECONDARY OUTCOMES:
Identifying Risk Factors for Insulin Resistance in each group | Baseline
  Information on each individual gathered regarding Lifestyle and Nutritional Habits including Social/Economic condition, Family History for obesity, diabetes and hypertension, perinatal history, early feeding and detailed Nutritional History; including sugar, carbohydrate and fat consumption, Physical activity, sleep quality, psychological stressors and performance at school. Data will be gathered for each group; Insulin Resistant and Non-Insulin resistance to determine associations between the two.

REFERENCES:
- [Background] Ighbariya A, Weiss R. Insulin Resistance, Prediabetes, Metabolic Syndrome: What Should Every Pediatrician Know? J Clin Res Pediatr Endocrinol. 2017 Dec 30;9(Suppl 2):49-57. doi: 10.4274/jcrpe.2017.S005. Epub 2017 Dec 27. PMID 29280741
- [Background] Lobstein T, Jackson-Leach R, Moodie ML, Hall KD, Gortmaker SL, Swinburn BA, James WP, Wang Y, McPherson K. Child and adolescent obesity: part of a bigger picture. Lancet. 2015 Jun 20;385(9986):2510-20. doi: 10.1016/S0140-6736(14)61746-3. Epub 2015 Feb 19. PMID 25703114
- [Background] de Onis M, Blossner M, Borghi E. Global prevalence and trends of overweight and obesity among preschool children. Am J Clin Nutr. 2010 Nov;92(5):1257-64. doi: 10.3945/ajcn.2010.29786. Epub 2010 Sep 22. PMID 20861173
- [Background] Kelly AS, Barlow SE, Rao G, Inge TH, Hayman LL, Steinberger J, Urbina EM, Ewing LJ, Daniels SR; American Heart Association Atherosclerosis, Hypertension, and Obesity in the Young Committee of the Council on Cardiovascular Disease in the Young, Council on Nutrition, Physical Activity and Metabolism, and Council on Clinical Cardiology. Severe obesity in children and adolescents: identification, associated health risks, and treatment approaches: a scientific statement from the American Heart Association. Circulation. 2013 Oct 8;128(15):1689-712. doi: 10.1161/CIR.0b013e3182a5cfb3. Epub 2013 Sep 9. PMID 24016455
- [Background] Govers E. Obesity and Insulin Resistance Are the Central Issues in Prevention of and Care for Comorbidities. Healthcare (Basel). 2015 Jun 4;3(2):408-16. doi: 10.3390/healthcare3020408. PMID 27417770
- [Background] Kahn SE, Hull RL, Utzschneider KM. Mechanisms linking obesity to insulin resistance and type 2 diabetes. Nature. 2006 Dec 14;444(7121):840-6. doi: 10.1038/nature05482. PMID 17167471
- [Background] Levy-Marchal C, Arslanian S, Cutfield W, Sinaiko A, Druet C, Marcovecchio ML, Chiarelli F; ESPE-LWPES-ISPAD-APPES-APEG-SLEP-JSPE; Insulin Resistance in Children Consensus Conference Group. Insulin resistance in children: consensus, perspective, and future directions. J Clin Endocrinol Metab. 2010 Dec;95(12):5189-98. doi: 10.1210/jc.2010-1047. Epub 2010 Sep 8. PMID 20829185
- [Background] Kurtoglu S, Hatipoglu N, Mazicioglu M, Kendirici M, Keskin M, Kondolot M. Insulin resistance in obese children and adolescents: HOMA-IR cut-off levels in the prepubertal and pubertal periods. J Clin Res Pediatr Endocrinol. 2010;2(3):100-6. doi: 10.4274/jcrpe.v2i3.100. Epub 2010 Aug 2. PMID 21274322
- [Background] van der Aa MP, Fazeli Farsani S, Knibbe CA, de Boer A, van der Vorst MM. Population-Based Studies on the Epidemiology of Insulin Resistance in Children. J Diabetes Res. 2015;2015:362375. doi: 10.1155/2015/362375. Epub 2015 Jul 27. PMID 26273668
- [Background] van der Aa MP, Knibbe CA, Boer A, van der Vorst MM. Definition of insulin resistance affects prevalence rate in pediatric patients: a systematic review and call for consensus. J Pediatr Endocrinol Metab. 2017 Feb 1;30(2):123-131. doi: 10.1515/jpem-2016-0242. PMID 27984205
- [Background] Goran MI, Gower BA. Longitudinal study on pubertal insulin resistance. Diabetes. 2001 Nov;50(11):2444-50. doi: 10.2337/diabetes.50.11.2444. PMID 11679420
- [Background] Moran A, Jacobs DR Jr, Steinberger J, Hong CP, Prineas R, Luepker R, Sinaiko AR. Insulin resistance during puberty: results from clamp studies in 357 children. Diabetes. 1999 Oct;48(10):2039-44. doi: 10.2337/diabetes.48.10.2039. PMID 10512371
- [Background] Ling JC, Mohamed MN, Jalaludin MY, Rampal S, Zaharan NL, Mohamed Z. Determinants of High Fasting Insulin and Insulin Resistance Among Overweight/Obese Adolescents. Sci Rep. 2016 Nov 8;6:36270. doi: 10.1038/srep36270. PMID 27824069
- [Background] van der Aa MP, Fazeli Farsani S, Kromwijk LA, de Boer A, Knibbe CA, van der Vorst MM. How to screen obese children at risk for type 2 diabetes mellitus? Clin Pediatr (Phila). 2014 Apr;53(4):337-42. doi: 10.1177/0009922813509480. Epub 2013 Nov 14. PMID 24243989